CLINICAL TRIAL: NCT05188911
Title: Analysis of Next Generation PET and Liquid Biopsy to Monitor mCRPC Treated With Abiraterone: ANGELA Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Dr., Fudan University
Other Study IDs: ANGELA trial
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — abiraterone; Prednisone; Androgen Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mCRPC: Patients would be treated with 1000mg abiraterone qd. Patients would be treated with 5mg prednisone bid. Patients would get medical or surgical castration.
  Interventions: Drug: Abiraterone; Drug: Prednisone; Drug: Androgen deprivation therapy

INTERVENTIONS:
Drug: Abiraterone — Patients would be treated with 1000mg abiraterone qd.
Drug: Prednisone — Patients would be treated with 5mg prednisone bid.
Drug: Androgen deprivation therapy — Patients would get medical or surgical castration.

SUMMARY:
By incorporating dual-tracer PET/CT (PSMA and FDG) and ctDNA, we aimed to evaluate lesion heterogeneity and genomic change of mCRPC patients receiving novel hormonal therapy. The relationship between treatment response and different molecular characterization, as well as imaging features would also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as mCRPC according to EAU-ESTRO-SIOG 2016 and PSA > 10ng/ml;
2. No previous treatment with novel hormonal therapy;
3. ECOG 0-2;
4. Normal organ function, WBC >= 3000/mm3 or Neutrophil >= 1500/mm3;
5. Aged 18 to 85 years old when issuing written informed consent;
6. Life expectancy > 12 months.
7. Consent and able to carry out follow-up visit and cooperate with all other study procedures.

Exclusion Criteria:

1. Severe disease or other medical conditions suggesting a high risk of death within 1 year, which may interfere with follow-up. Decided by investigator;
2. Diagnosed with any other malignant tumor within 3 years before enrollment;
3. Unable to provide necessary follow-up information;
4. Other conditions that are judged as ineligible by the investigator.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic castration-resistant prostate cancer
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Lesion heterogeneity on dual-tracer PET/CT | 90 days
Genomic change | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pan J, Wu J, Wang B, Zhu B, Liu X, Gan H, Wei Y, Jin S, Hu X, Wang Q, Song S, Liu C, Ye D, Zhu Y. Interlesional response heterogeneity is associated with the prognosis of abiraterone treatment in metastatic castration-resistant prostate cancer. Med. 2024 Dec 13;5(12):1475-1484.e3. doi: 10.1016/j.medj.2024.07.020. Epub 2024 Aug 15. PMID 39151419